CLINICAL TRIAL: NCT05499494
Title: Clinical Evaluation of Bioactive Injectable Resin Composite Versus Conventional Nanohybrid Composite in Posterior Restorations, 18 m Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of Bioactive Injectable Resin Composite in Posterior Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hazem Mohamed El Deriny, Assistant lecturer at operative dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Injectable resin composite
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Dental Restoration Failure
Keywords: Injectable composite; Nano hybrid composite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- injectable composite (Experimental): The material will be applied according to manufacturer instructions. BEAUTIFIL Flow Plus X will be applied directly into the cavity and create the shape desired in layers not exceeding 2 mm, and light cured for 20 seconds.
  Interventions: Other: Beautifil Flow Plus X F00 injectable composite
- Nanohybrid resin composite (Active Comparator): The nanohybrid resin composite will be applied to the the cavity using the conventional incremental technique according to manufacturer instructions.
  Interventions: Other: Tetric N ceram resin composite

INTERVENTIONS:
Other: Beautifil Flow Plus X F00 injectable composite — bioactive injectable composite
  Arms: injectable composite
Other: Tetric N ceram resin composite — Nano hybrid resin composite
  Arms: Nanohybrid resin composite

SUMMARY:
The aim of the study is to evaluate the clinical performance of new bioactive injectable composite compared to nanohybrid composite during the restoration of posterior cavities

DETAILED DESCRIPTION:
Statement of the problem:

Marginal defects of composite fillings are often thought to be caused by poor adaptation of the restorative material to the cavity wall. To avoid these defects, particularly in posterior teeth, the use of flowable composites has been advocated because of their ability to 'wet' and adapt well to cavity margins and walls. However, flowable composites have a lower filler content and usually weaker mechanical properties than conventional composites.

The continued development of resin composites has led to formulations designed to further simplify the filling procedure, provide better mechanical properties, reduce the effect of polymerization shrinkage stresses and improve aesthetics. Recently, a new type of highly filled flowable composite has been developed. It is characterized by its high viscosity and is claimed to have improved mechanical properties not dissimilar from conventional composite restorative materials. This composite contains nano-sized filler particles, and due to its consistency, the material has been referred to as an 'injectable composite'.

Rationale for carrying out the trial:

The rationale of this study is to evaluate the mechanical performance of injectable composite resin against nanohybrid composites, because of its easy handling, time-saving, better margin adaptation, and the gain of extra mechanical properties at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Participants:

  1. Age range 20-50 years.
  2. Males Or females .
  3. Co-operative patients approving to participate in the trial.
* Teeth:

  1. class I or II carious lesions premolars and molars.
  2. Vital upper or lower teeth with no signs of irreversible pulpitis and pulpal necrosis.
  3. Presence of favorable occlusion and teeth are in normal contact with the adjacent teeth.

Exclusion Criteria:

* Participants:

  1. Patients with general systemic illness.
  2. Allergic history against any component of used material.
  3. Disabilities.
  4. Pregnancy
  5. Xerostomia.
  6. Lack of compliance.
  7. Evidence of parafunctional habits.
  8. Temporomandibular joint disorders.
* Teeth:

  1. Periapical pathology or signs of pulpal pathology.
  2. Endodontically treated teeth.
  3. Tooth hypersensitivity.
  4. Possible prosthodontic restoration of teeth.
  5. Heavy occlusion and occlusal contacts or history of bruxism.
  6. Severe periodontal affection.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in the clinical performance | From baseline to 18 months
  Measured using modified USPHS criteria

CONTACTS AND LOCATIONS:
Overall Officials: Mai Mamdouh, PhD, Study Director — Cairo University
Locations (1):
- Faculty of dentistry, Cairo University, Cairo, Egypt